CLINICAL TRIAL: NCT03252808
Title: Phase I Study of Combination with TBI-1401(HF10), a Replication-competent HSV-1 Oncolytic Virus, and Chemotherapy in Patients with Stage III or IV Unresectable Pancreatic Cancer.
Brief Title: Phase I Study of TBI-1401(HF10) Plus Chemotherapy in Patients with Unresectable Pancreatic Cancer.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBI1401-03
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer Stage III; Pancreatic Cancer Stage IV
Keywords: Unresectable pancreatic cancer; Metastatic pancreatic cancer; Pancreatic adenocarcinoma; TBI-1401(HF10); HF10; Oncolytic virus; Oncolytic viral immunotherapy; Gemcitabine; Nab-paclitaxel; Albumin-bound paclitaxel; Abraxane; Tegafur-gimeracil-oteracil potassium; TS-1; canerpaturev
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TBI-1401(HF10) + Gem/nab-PTX (Experimental): 1x10^6 or 1x10^7 TCID50/mL TBI-1401(HF10) administered to the tumor in a total volume up to 2.0 mL (injection volume will be adjusted based on the tumor size) by EUS-guided intratumoral injection and 1000 mg/m^2 Gemcitabine and 125 mg/m^2 Nab-paclitaxel injected by intravenous infusions.
  Interventions: Biological: TBI-1401(HF10); Drug: Gemcitabine; Drug: Nab-paclitaxel
- TBI-1401(HF10) + TS-1 (primary) (Experimental): 1x10^6 or 1x10^7 TCID50/mL TBI-1401(HF10) administered to the primary tumor in a total volume up to 2.0 mL (injection volume will be adjusted based on the tumor size) by EUS-guided intratumoral injection and TS-1 administered by oral.
  Interventions: Biological: TBI-1401(HF10); Drug: TS-1
- TBI-1401(HF10) + TS-1 (primary and meta) (Experimental): 1x10^6 or 1x10^7 TCID50/mL TBI-1401(HF10) administered to the primary tumor in a total volume up to 2.0 mL (injection volume will be adjusted based on the tumor size) by EUS-guided intratumoral injection and hepatic metastasis in a total volume up to 2.0 mL (injection volume will be adjusted based on the tumor size) by EUS-guided intratumoral injection or percutaneous injection and TS-1 administered by oral.
  Interventions: Biological: TBI-1401(HF10); Drug: TS-1

INTERVENTIONS:
Biological: TBI-1401(HF10) — 1x10^6 or 1x10^7 TCID50/mL TBI-1401(HF10) administered by intratumoral injection at 2-week intervals. Patients may continue to receive the injections for up to 1 year if eligible for injection.
  Other Names: HF10; canerpaturev
Drug: Gemcitabine — 1000 mg/m^2 Gemcitabine administered by intravenous infusion at weekly for 3 weeks followed by a week of rest.
  Other Names: Gemzar
  Arms: TBI-1401(HF10) + Gem/nab-PTX
Drug: Nab-paclitaxel — 125 mg/m^2 Nab-paclitaxel administered by intravenous infusion at weekly for 3 weeks followed by a week of rest.
  Other Names: Abraxane
  Arms: TBI-1401(HF10) + Gem/nab-PTX
Drug: TS-1 — TS-1 (40-60 mg per body surface area) administered by oral at twice daily for 4 weeks followed by 2 weeks of rest.
  Other Names: Tegafur-gimeracil-oteracil potassium
  Arms: TBI-1401(HF10) + TS-1 (primary and meta); TBI-1401(HF10) + TS-1 (primary)

SUMMARY:
The purpose of this study is to determine the recommended dose of TBI-1401(HF10) treatment in combination with chemotherapy (Gemcitabine + Nab-paclitaxel or TS-1) in patients with stage III or IV unresectable pancreatic cancer.

DETAILED DESCRIPTION:
A Phase I, open-label, multi-center study to determine the recommended dose of TBI-1401(HF10) treatment in combination with chemotherapy (Gemcitabine + Nab-paclitaxel or TS-1) in patients with stage III or IV unresectable pancreatic cancer. Patients with stage IV must failed a gemcitabine based first-line chemotherapy.

Patients with stage III will receive the repeated intratumoral injection of TBI-1401(HF10) at recommended dose at 2-week intervals in combination with intravenous infusion of 1000 mg/m^2 Gemcitabine and 125 mg/m^2 Nab-paclitaxel at weekly for 3 weeks followed by 1 week rest.

Patients with stage IV will receive the repeated intratumoral injection of TBI-1401(HF10) at recommended dose at 2-week intervals in combination with oral of 40 - 60 mg TS-1 at twice daily for 4 weeks followed by 2 weeks rest.

Patients will receive the combination therapy of TBI-1401(HF10) + chemo for up to 1 year if eligible for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed unresectable pancreatic cancer (stage III or IV) based on the General Rules for the Study of Pancreatic Cancer (The 7th edition), and never received anti-cancer therapy (radiation therapy, chemotherapy, immunotherapy, surgery, clinical trials).
* Patients with primary lesion will be intratumorally injectable for TBI-1401(HF10) by EUS (endoscopic ultrasound).
* Patients must be ≧20 years of age.
* Patients must have at least one measurable lesion evaluated by Computed Tomography (CT) scan on RECIST ver.1.1 at pre-treatment.
* Patients must have a life expectancy ≧12 weeks.
* Patients must have an ECOG PS (Eastern Cooperative Oncology Group Performance Status) of 0-1.
* Patients demonstrated adequate organ function (≦7 days prior to treatment).
* Females of childbearing potential must have a negative urine or serum pregnancy test within 1 week prior to start of treatment.
* Patients must be able to understand the study and willing to sign a written informed consent document.

Exclusion Criteria:

* Patients receiving anti-herpes medication within 1 week prior to TBI-1401(HF10) treatment (except local treatment such as ointment).
* Patients with a significant tumor bleeding or coagulation abnormality that could not treat intratumoral injection or biopsy in safe.
* Patients with clinically evident Hepatitis B surface antigen (HBs) positive, Hepatitis C virus (HCV) antibody positive and HSV-RNA positive, Human Immunodeficiency Virus (HIV) antibody positive.
* Patients with the active symptom of Epstein-Barr virus (EBV) infection.
* Patients with active CNS metastases.
* Patients with ascites, except acceptable mild ascites.
* Patients with multiple cancer.
* Patients need to treat anticoagulant or antiplatelet agent.
* Patients has a history of allergy for CT contrast agent, live vaccine, any drug excipients, Nab-paclitaxel, Gemcitabine, or any study drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2035-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Through 1st TBI-1401(HF10) injection to before 3rd injection (basically 4 weeks).
  Determine the recommended dose of TBI-1401(HF10) in combination with Gemcitabine and Nab-paclitaxel.

SECONDARY OUTCOMES:
Adverse Events (AEs) | Through 1st TBI-1401(HF10) injection to study completion (up to 13 month).
  Evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE version 4.0).
Objective response rate (ORR) by RECIST | At 16 weeks and through study completion (up to 1 year).
  Overall tumor response evaluated by RECIST version 1.1
Objective response rate (ORR) by irRECIST | At 16 weeks and through study completion (up to 1 year).
  Overall tumor response evaluated by irRECIST.
Progression-free survival (PFS) by RECIST | Through disease progression (up to 1 year).
  Evaluation the time to progression during and after the treatment.
Progression-free survival (PFS) by irRECIST | Through disease progression (up to 1 year).
  Evaluation the time to progression during and after the treatment.

OTHER OUTCOMES:
Overall survival (OS) | From 1st treatment to death (up to 2 years).
  Evaluation the overall survival.
1 year survival rate | for 1 year.
  Determine the 1 year survival rate of patient who received treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Takara Bio Inc., Study Director — Clinical Development & Strategy Division 2
Locations (8):
- Japan (8):
  - Clinical Site, Nagoya, Aichi-ken
  - Clinical Site, Chiba, Chiba
  - Clinical Site, Kashiwa, Chiba
  - Clinical Site, Yokohama, Kanagawa
  - Clinical Site, Osaka, Osaka
  - Clinical Site, Chūōku, Tokyo
  - Clinical Site, Koto-Ku, Tokyo
  - Clinical Site, Nagoya

IPD SHARING:
Plan to Share IPD: No